CLINICAL TRIAL: NCT06353035
Title: Biodiversity Interventions for Well-being, Neighborhood Rewilding
Brief Title: Biodiversity Interventions for Well-Being
Acronym: BIWE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Resources Institute Finland (Other Government)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NaturalResourcesIFinland; 346136 (Other Grant/Funding Number: Strategic Research Council Finland); 346138 (Other Grant/Funding Number: Strategic Research Council Finland)
Record Dates: First submitted 2024-03-27; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-03

CONDITIONS: Microbial Colonization; Immune System Diseases; Well-Being, Psychological; Nature, Human
Keywords: Commensal microbiome; Salivary cytokines; Planetary health; Well-being
MeSH Terms: conditions — Communicable Diseases; Immune System Diseases; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Intervention-control study in which intervention study subjects private yards are rewilded and control receives no treatment.
Masking Description: The research subjects were not randomized or masked to the intervention and control group, because the control group needs volunteers who have no intention of following the yard management instructions advised to the intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rewilding (Experimental): Private yards of the intervention study subjects will be modified with berry bushes, fruit trees, perennial yard plants, meadow flowers, cultivation boxes, organic mulch materials, decaying deadwood, leaf compost and organic plant growing media with high microbial diversity.
  Interventions: Other: Rewilding
- Control (No Intervention): The control group's yards will not be modified. Control group receives inorganic fertilizers, moss remover and ant control insecticide (Myrr®; active ingredient imidacloprid 0.03 % w/w).

INTERVENTIONS:
Other: Rewilding — Private yards of the intervention study subjects will be modified with vegetation and deadwood.
  Arms: Rewilding

SUMMARY:
Biodiversity is essential for nature and human well-being. Land use has reduced biodiversity in cities, which weakens the functionality of the urban ecosystems and the well-being of citizens. This may also increase the risk of immune-mediated disorders among urban dwellers.

In Biodiversity interventions for well-being (BIWE), microbial biodiversity interventions are performed to increase biodiversity in urban built areas. Results from the intervention trials are combined with publicly available land cover and ecological data. These are analyzed from the viewpoint of shifts in ecosystems and human well-being and immune regulation, ecological quality, and urban planning.

The investigators set up an intervention study in which urban private yards are rewilded with diverse vegetation and decaying deadwood and plant residuals. The investigators aim to evaluate the effect of rewilding, and yard management practices on commensal microbiome, cortisol levels and well-being and salivary cytokine levels, and gene pathways.

DETAILED DESCRIPTION:
Our specific aims are:

To assess if rewilding diversifies health-associated skin microbiota and is associated with salivary cytokine levels, gene pathways, cortisol levels and commensal microbiota.

Assess whether there are patterns in the microbiome associated with the salivary cytokine levels and hair cortisol levels.

Assess whether rewilding affects health and psychological measures, such as Perceived Stress Scale (PSS), Warwick-Edinburgh Mental Wellbeing Scale (SWEMWS), Depression Scale (DEPS) and Nature Relatedness Scale (NR6).

The investigators will recruit approximately 42 (21 study subjects per treatment) subjects living in a detached house or terraced house in urban areas and aged between 18-72.

The medical exclusion criteria include immunosuppressive medications, immune deficiencies, a disease affecting immune response (e.g., colitis ulcerosa, rheumatoid arthritis, Crohn's disease, diabetes), cancer diagnosis within the last year or on-going cancer treatment. Other exclusion criteria include incompetency and living outside city area.

ELIGIBILITY:
Inclusion Criteria:

* Living in a detached or terraced house in urban area

Exclusion Criteria:

* Immunosuppressive medications
* Immune deficiencies
* a disease affecting immune response (e.g., colitis ulcerosa, rheumatoid arthritis, Crohn's disease, diabetes)
* cancer diagnosis within the last year or on-going cancer treatment
* Incompetency
* Living outside city area.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Skin Gammaproteobacteria | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Difference on skin gammaproteobacterial diversity between rewilding and control group

SECONDARY OUTCOMES:
Salivary cytokines | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Interleukin-6 and -10 measured from saliva
Difference in diversity (Alpha and beta diversity) of skin, saliva and stool microbiota | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  It will be analyzed if microbial communities are different between treatments
Difference in observed species richness of skin, saliva and stool microbiota | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  It will be analyzed if microbial communities are different between treatments
Difference in taxonomies of skin, saliva and stool microbiota | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  It will be analyzed if microbial communities are different between treatments
Difference in microbial gene pathways of saliva and stool microbiota | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Will be analyzed with shotgun sequencing if gene pathways are different between treatments
Cortisol levels | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Cortisol levels measured from hair samples
Perceived Stress Scale | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Lower score on a perceived stress scale among intervention treatment compared to control that indicates lower perceived stress levels among intervention treatment. Minimum 0, maximum 40.
Warwick-Edinburgh Mental Wellbeing Scale | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Higher score on a Warwick-Edinburhg Mental Wellbeing scale among intervention treatment compared to control that indicates better mental well-being among intervention treatment. Minimum 14, maximum 70.
Depression Scale | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Lower score on a Depression scale among intervention treatment compared to control that indicates lower levels of depression symptoms among intervention treatment. Minimum 0, maximum 60.
Nature Relatedness Scale | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Higher score on a Nature Relatedness scale among intervention treatment compared to control that indicates stronger sense of connectedness to nature among intervention treatment. Minimum 6, maximum 30.
Metabolites in urine | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Metabolites of harmful substances are measured from the urine sample.

OTHER OUTCOMES:
Associations between environmental factors and microbial measurements, salivary cytokine levels, hair cortisol levels, perceived well-being | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  associations between environmental factors (vegetation, deadwood, and polypore richness, land cover categories and other yard characteristics), yard management practices, activities at the yard, salivary cytokine levels and bacterial measurements (diversity, and taxonomic and functional features).

CONTACTS AND LOCATIONS:
Overall Officials: Aki Sinkkonen, Principal Investigator — Natural Resources Institute Finland
Locations (1):
- Natural Resources Institute Finland, Helsinki, Uusimaa, Finland